CLINICAL TRIAL: NCT02118012
Title: Evaluation of Safety, Tolerability, and Antiviral Activity of Chlorcyclizine HCl Alone or in Combination With Ribavirin in Patients With Chronic Hepatitis C
Brief Title: Evaluation of Safety, Tolerability, and Antiviral Activity of Chlorcyclizine HCl in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140084; 14-DK-0084 (Other: NIDDK/NIH)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-09-17

CONDITIONS: Chronic Hepatitis C
Keywords: Chlorcyclizine HCL; Direct Acting Antivirals; Ribavirin; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — chlorcyclizine; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorcyclizine and RBV (Active Comparator): Chlorcyclizine HCl and Ribavirin
  Interventions: Drug: Chlorcyclizine HCl; Drug: Ribavirin
- Chlorcyclizine HCl only (Active Comparator): Chlorcyclizine HCl only
  Interventions: Drug: Chlorcyclizine HCl

INTERVENTIONS:
Drug: Chlorcyclizine HCl — Chlorcyclizine HCl (75 mg twice daily)
  Other Names: CCZ
Drug: Ribavirin — RBV was dosed via a weight-based regimen of 1000 mg daily<75 kg and 1200 mg daily ≥75 kg.
  Other Names: RBV
  Arms: Chlorcyclizine and RBV

SUMMARY:
Background:

- Hepatitis C is a liver disease caused by the hepatitis C virus. It is the most common cause of serious liver disease in the United States. Many people have few if any symptoms. It can lead to cirrhosis, which can cause liver failure and cancer. Researchers want to study how a medicine called chlorcyclizine works in patients with hepatitis C. They want to see if it can be used to treat hepatitis C alone or when used with the standard hepatitis C treatment drug ribavirin.

Objectives:

- To see if chlorcyclizine can be used to treat hepatitis C alone or in combination with the drug ribavirin.

Eligibility:

- Adults with chronic hepatitis C who either have never been treated for it or have relapsed after prior treatment.

Design:

* Participants will be screened with medical history, physical exam, blood and urine tests, and a questionnaire. They will also have an ultrasound of their abdomen and electrocardiogram. Some of these tests will be repeated throughout the study.
* Participants will spend 3 days as an inpatient to be monitored while starting study drug. They will be assigned randomly to a group and will begin taking the study drug. Blood will be taken frequently.
* Group I will take the study drug twice a day for 28 days.
* Group II will take the study drug twice a day and ribavirin twice a day for 28 days.
* Participants will visit the clinic every 7 days for 28 days.
* After participants stop taking the study drug, they will have 5 follow-up visits over 3 months.

DETAILED DESCRIPTION:
Up to 50 patients with chronic hepatitis C, who are treatment na(SqrRoot) ve or relapsers to any interferon/ribavirin regimen will be enrolled into this pilot study evaluating chlorcyclizine HCl with or without ribavirin (RBV) as antiviral therapy. Adult patients (greater than or equal to18 years of age) with evidence of active chronic hepatitis C infection (all genotypes) with detectable HCV RNA in serum >10,000 IU/mL without contraindications to chlorcyclizine HCl or ribavirin or evidence/history of hepatic decompensation will be enrolled. Patients will be monitored for at least two months with regular testing for ALT and HCV RNA quantitative levels before treatment and will undergo admission to start therapy, which includes a thorough medical evaluation and timed blood sampling. Patients will be randomized to one of two treatment groups; one with chlorcyclizine HCl (75 mg twice daily) and the other with RBV+ chlorcyclizine HCl (75 mg twice daily). For all genotypes, RBV will be dosed based on weight (1000 mg daily <75 kg and 1200 mg daily greater than or equal to 75 kg). At each clinic visit, patients will be questioned about side effects and symptoms, undergo a focused physical examination, and have blood taken for complete blood counts, HCV RNA, PT/INR and routine liver tests (ALT, AST, alkaline phosphatase, direct and total bilirubin, and albumin). At the end of 28 days of treatment, patients will undergo a repeat thorough medical evaluation inclusive of a complete physical exam, symptom scale evaluation, complete blood counts, routine liver tests, and HCV serology panels. The primary endpoint of therapy will be a decline in quantitative HCV RNA viral levels after 28 days of treatment as compared to baseline viral titers and between groups. Several secondary endpoints will be measured, including side effects of therapy, ALT levels, quantification of chlorcyclizine HCl and its metabolites in serum, and quality of life. Therapy will be stopped for intolerance to RBV and/or chlorcyclizine HCl (which will be carefully defined).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults, ages 18 and above;
* Chronic hepatitis C (HCV RNA in serum for more than 6 months);
* HCV RNA in serum at or above 10,000 IU/mL;
* Treatment naive patients defined as individuals whom have never undergone any form of interferon and ribavirin therapy for chronic HCV infection or relapsers defined as reappearance of HCV RNA in serum after treatment (with any form of interferon and ribavirin therapy) was discontinued and an end-of-treatment response was achieved;
* No major contraindications to agents being used (chlorcyclizine HCl and ribavirin);
* Females of childbearing potential must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours before the first dose of study drug;
* Women of childbearing potential and men, participants and partners, must use highly effective methods of birth control to minimize the risk of pregnancy and must follow instructions for birth control for the entire duration of the study including a minimum of 24 weeks after the last dose of ribavirin. Two forms of birth control are required from the time of screening throughout the duration of the on-treatment study period and for at least 24 weeks after the last dose of ribavirin. Examples of effective birth control include: condom with spermicide; diaphragm with spermicide; cervical cap with spermicide; female condom; intrauterine devices (IUDs); vasectomy in men;

EXCLUSION CRITERIA:

* Liver or any other organ transplant (including hematopoietic stem cell transplants) other than cornea and hair;
* Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment;
* Documented or suspected HCC, as evidenced by previously obtained imaging studies or liver biopsy (or on a screening imaging study/liver biopsy if this was performed);
* Evidence of decompensated liver disease including, but not limited to, bilirubin >4 mg/dL, albumin <3.0 gm/dL, prothrombin time >2 sec prolonged or a history or presence of ascites, bleeding varices, or hepatic encephalopathy. Patients with ALT levels >500 U/L will not be enrolled but may be followed until three determinations are below this level;
* Evidence of a medical condition contributing to chronic liver disease other than chronic HCV infection (such as, but not limited to: acute hepatitis C infection, hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures);
* History of chronic hepatitis B virus (HBV) as documented by HBV serologies (eg, HBsAg-seropositive). Subjects with resolved HBV infection may participate (eg, HBsAb-seropositive with concurrent HBsAg-seronegative);
* Any prior exposure to direct-acting antiviral therapies for chronic HCV infection;
* History of HIV infection;
* History of hemoglobinopathies (eg. thalassemia major or sickle cell anemia), diagnoses associated with an increased baseline risk for anemia (eg, spherocytosis), hemolytic anemia, or diseases in which anemia would be medically problematic, or hemophilia;
* Confirmed, uncontrolled hypertension (any screening systolic blood pressure greater than or equal to 160 mmHg or diastolic blood pressure greater than or equal to 100 mmHg should be excluded unless discussed with the central medical monitor);
* Any other medical and/or social reason, including active substance abuse as defined by DSM-IV, Diagnostic Criteria for Drug and Alcohol Abuse, which in the opinion of the investigator would make the candidate inappropriate for participation in this study;
* Significant systemic or major illnesses other than liver disease, including, but not limited to, clinically significant emphysema or chronic bronchitis, symptomatic benign prostatic hypertrophy, glaucoma, gastrointestinal motility related illnesses, congestive heart failure, renal failure (eGFR <50 mL/min), and active coronary artery disease;
* Significant prior history suggestive of cardiovascular instability, including but not limited to evidence of significant myocardial ischemia, unstable re-entry phenomena, other significant dysrhythmias and/or uncontrolled hypertension;
* Inability to tolerate oral medication;
* For relapsers: exposure to interferon based therapy with ribavirin within 12 weeks prior to screening;
* Allergy or hypersensitivity to chlorcyclizine HCl or ribavirin;
* Any known contraindication to ribavirin, not otherwise specified;
* Inability to refrain from operating heavy machinery while on therapy;
* Breastfeeding women;
* Inability to understand or sign informed consent;
* Active use of chlorcyclizine HCl or another piperazine class antihistamine within 6 months of enrollment;
* Inability to abstain from piperazine class antihistamines during enrollment in the clinical trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03-20; Primary Completion 2014-03-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Koh, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Koh C, Dubey P, Han MAT, Walter PJ, Garraffo HM, Surana P, Southall NT, Borochov N, Uprichard SL, Cotler SJ, Etzion O, Heller T, Dahari H, Liang TJ. A randomized, proof-of-concept clinical trial on repurposing chlorcyclizine for the treatment of chronic hepatitis C. Antiviral Res. 2019 Mar;163:149-155. doi: 10.1016/j.antiviral.2019.01.017. Epub 2019 Jan 31. PMID 30711416
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-DK-0084.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorcyclizine and RBV: Chlorcyclizine HCl and Ribavirin
  Chlorcyclizine HCL plus Ribavirin: RBV+ chlorcyclizine HCl (75 mg twice daily)
- Chlorcyclizine HCl Only: chlorcyclizine HCl (75 mg twice daily)
  Chlorcyclizine HCL Only: chlorcyclizine HCl (75 mg twice daily)
Period: Overall Study
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only
Started | 12 | 12
Day 5 | 12 | 11
Day 14 | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [47 to 60] | 57 [54 to 61] | 56 [50 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HCV Genotype [Count of Participants; unit: Participants]
  1A | 7 | 4 | 11
  1B | 3 | 4 | 7
  2 | 0 | 1 | 1
  3 | 1 | 2 | 3
  4 | 0 | 1 | 1
  6 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum HCV RNA Viral Titer From Baseline to 28 Days
Time Frame: Baseline and 28 days
Measure: Median (Inter-Quartile Range); unit: log IU/ml
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only
Number analyzed (Participants) | 12 | 10
log IU/ml | -0.46 [-0.83 to -0.04] | -0.11 [-0.21 to 0.21]

2. Primary Outcome: Number of Participants Who Tolerated the Drug at the Prescribed Dose for the Duration of Therapy
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only
Number analyzed (Participants) | 12 | 12
Participants | 12 | 11

3. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels From Baseline to 28 Days
Time Frame: Baseline and 28 days
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only
Number analyzed (Participants) | 12 | 10
U/L | 26 [5.75 to 45.25] | 6 [0.5 to 15]

4. Secondary Outcome: Maximum Chlorcyclizine HCL Weeks 1-4
Description: Chlorcyclizine HCL concentration was measured once a week in the morning. This outcome is the maximum over the four weeks.
Time Frame: Weeks 1-4
Population: Concentration measurements were not available for 1 Chlorcyclizine and RBV participant and for the 2 Chlorcyclizine HCl only participants who withdrew from the study
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only
Number analyzed (Participants) | 11 | 10
ng/ml | 211 [125 to 240] | 251 [153 to 285]

ADVERSE EVENTS:
Time Frame: 28 days
Description: Monitoring of adverse events was performed from the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 with modification for patients with liver disease.
Arm/Group | Chlorcyclizine and RBV | Chlorcyclizine HCl Only
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorcyclizine and RBV (N=12) | Chlorcyclizine HCl Only (N=12)
Drowsiness (General disorders) | 6 | 5
Dry Mouth (Gastrointestinal disorders) | 9 | 10
Light Headedness (General disorders) | 2 | 4
Nervousness (Nervous system disorders) | 6 | 2
Inability to concentrate (Psychiatric disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 0
Headaches (Nervous system disorders) | 2 | 2
Numbness or Tingling (Nervous system disorders) | 2 | 3
Difficulty Urinating (Renal and urinary disorders) | 2 | 1
Fatigue (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02118012/Prot_SAP_000.pdf